CLINICAL TRIAL: NCT05737667
Title: Advancing mHealth-supported Adoption and Sustainment of an Evidence-based Mental Health Intervention for Youth in a School-based Delivery Setting in Sierra Leone
Brief Title: Advancing mHealth-supported Adoption and Sustainment of an Evidence-based Mental Health Intervention in Sierra Leone
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022003442; R01MH130320 (NIH)
Record Dates: First submitted 2023-02-02; First posted 2023-02-21 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- YRI+Mobile Supervision (Experimental): Youth Readiness Intervention delivered by teachers receiving mobile-based supervision
  Interventions: Behavioral: Youth Readiness Intervention (YRI)
- YRI+Standard Supervision (Active Comparator): Youth Readiness Intervention delivered by teachers receiving standard supervision
  Interventions: Behavioral: Youth Readiness Intervention (YRI)
- Control (No Intervention): Wait listed control

INTERVENTIONS:
Behavioral: Youth Readiness Intervention (YRI) — The YRI is a culturally adapted group intervention that integrates common practice elements of cognitive behavioral and interpersonal therapies. The YRI's core treatment elements target improving emotion regulation skills, interpersonal functioning, and problem-solving skills. The YRI has 12 session that last about 90 minutes. The YRI will be delivered in schools by teachers receiving either mobile-based supervision or standard, in-person supervision.
  Arms: YRI+Mobile Supervision; YRI+Standard Supervision

SUMMARY:
This study will examine a new implementation strategy for the Youth Readiness Intervention (YRI), an evidence-based mental health intervention. The strategy will (a) leverage a delivery setting (schools) and workforce (teachers) used effectively in low- and middle- income countries; and (b) innovate with technology and mHealth tools to enhance mental health service delivery quality. The YRI will be implemented as an extracurricular resilience-building after school activity in Sierra Leone. Teachers will deliver the YRI and receive either mobile phone-supported supervision or standard in-person supervision. Mobile-based supervision will integrate WhatsApp, a free cross-platform messaging and voice service used widely throughout Africa, with mHealth digital tools. The mHealth tools will support supervision through key features, including voice activated content, fillable forms (i.e., YRI fidelity checklist), and visual dashboards to monitor fidelity. A hybrid type 3 implementation-effectiveness design will allow for evaluation of both mobile phone-based supervision as a new implementation strategy, and clinical effectiveness of the YRI on youth mental and behavioral health as secondary outcomes.

DETAILED DESCRIPTION:
This study will examine a new implementation strategy for the Youth Readiness Intervention (YRI), an evidence-based mental health intervention. The strategy will (a) leverage a delivery setting (schools) and workforce (teachers) used effectively in low- and middle- income countries; and (b) innovate with technology and mHealth tools to enhance mental health service delivery quality. The YRI will be implemented as an extracurricular resilience-building after school activity in Sierra Leone. Teachers will deliver the YRI and receive either mobile phone-supported supervision or standard in-person supervision. Mobile-based supervision will integrate WhatsApp, a free cross-platform messaging and voice service used widely throughout Africa, with new mobile-based digital tools. The mHealth tools will support supervision through key features, including voice activated content, fillable forms (i.e., YRI fidelity checklist), visual dashboards to monitor fidelity, and training videos to support school-based YRI delivery.

The Exploration, Preparation, Implementation, Sustainment framework, a broad multilevel, context-sensitive implementation science model, will guide the study. A hybrid type 3 implementation-effectiveness design will allow for evaluation of both mobile phone-based supervision as a new implementation strategy, and clinical effectiveness of the YRI on youth mental and behavioral health as secondary outcomes.

Aim 1 (Exploration and Preparation) will investigate barriers and facilitators to successful YRI implementation aided by mobile-based tools in Sierra Leone's secondary schools. A mixed methods evaluation with teachers, principals, and government ministry officials will inform co-development of an implementation blueprint prior to YRI delivery. User-centered design methods will be used to adapt the mHealth supervision app and incorporate WhatsApp to create an integrated user model of mobile phone-based supervision. Aim 2 (Implementation) will examine the feasibility, acceptability, cost, and fidelity to the YRI delivered by teachers receiving mobile-based supervision compared with those receiving standard supervision via a mixed methods approach. Aim 3 (Impact of Delivery Approach on YRI Effectiveness) will compare the effectiveness of the YRI in improving mental health, emotion regulation and daily functioning in youth (aged 14-24) when delivered in school settings by teachers who receive either mobile-based supervision (N=480 youth) or those who receive standard supervision (N=480 youth). Aim 4 (Sustainment) will (a) investigate mechanisms of adoption and sustainment of the YRI delivered by teachers through a mixed methods evaluation with teachers, youth, and principals; and (b) conduct a cost-effectiveness and return on investment analysis to evaluate relative costs vs. benefits of the YRI from a broad societal perspective, including educational outcomes.

ELIGIBILITY:
School Inclusion Criteria:

* We will include secondary schools in the Western Region that are willing to provide the Youth Readiness Intervention (YRI) as an extracurricular activity

School Exclusion Criteria:

* We will exclude schools that do not meet the inclusion criteria.

Teacher Inclusion Criteria:

* We will include teachers who are (a) currently employed at a Western Region urban or rural secondary school; (b) willing to provide the YRI as an extracurricular activity

Teacher Exclusion Criteria:

* We will exclude teachers who do meet inclusion criteria.

Youth Inclusion Criteria:

* We will include youth who are (a) currently enrolled in a secondary school in the Western Region (urban or rural); (b) male or female aged 14-24; (c) able to attend after school activities. We will require both youth assent and parental consent for all youth under age 18.

Youth Exclusion Criteria:

* We will exclude youth who do not meet all inclusion criteria and/or who report active, severe suicidality or psychosis as determined by a study social worker.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1454 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Fidelity | For 12 weeks, starting from the date of the first YRI session
  Fidelity will be measured with the YRI Fidelity Checklist, a tool developed and tested in previous trials that is completed after each YRI session.
Acceptability | An average of 24 weeks
  Acceptability, or the level of satisfaction with the intervention, will be assessed with the Johns Hopkins University Implementation Science Questionnaire. The scale has 12 items scored on a 4-point Likert scale: 1=Not at all, 2=A little bit, 3=A moderate amount, 4=A lot. Higher scores mean greater acceptability.
Appropriateness | An average of 24 weeks
  Appropriateness, or the relevance and fit of the intervention, will be assessed with Johns Hopkins University Implementation Science Questionnaire. The scale has 12 items scored on a 4-point Likert scale: 1=Not at all, 2=A little bit, 3=A moderate amount, 4=A lot. Higher scores mean greater appropriateness.

SECONDARY OUTCOMES:
emotion regulation skills | An average of 24 weeks
  Emotion regulation skills, or the ability to modulate emotional responses, will be measured with the Difficulties in Emotion Regulation Scale. This is a 36-item scale and responses are scored on a 5-point Likert scale: 1=Almost Never, 2=Sometimes, 3=About half the time, 4=Most of the time, 5=Almost always. Higher scores indicate poorer emotion regulation skills.
Anxiety and Depression | An average of 24 weeks
  Anxiety and Depression will be measured with the Hopkins Symptom Checklist, a 25-item inventory that measures symptoms of anxiety and depression. Part I of the measure has 10 items assessing anxiety symptoms and Part II has 15 items assessing depression symptoms. Each item is rated on a 4-point scale: 1 = Not at all, 2 = A little, 3 = Quite a bit, and 4 = Extremely. Item scores are summed to derive scores for the total scale and subscales, i.e., anxiety and depression. Higher scores reflect worse functioning.
Functional Impairment | An average of 1 year
  Functional Impairment will be measured by the World Health Organization Disability Assessment Schedule short-form. This scale contains 12 items and assesses functioning across five domains: mobility, self-care, understanding and communication, life activities and societal participation. Items are scored on a 5-point Likert scale (0-4) and summed to derive a total scale. Higher scores reflect worse functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Alethea Desrosiers, Ph.D., Principal Investigator — Brown University
Locations (1):
- Innovations for Poverty Action, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: Yes
The PI and her collaborators will abide by the principles for sharing research resources and data, as described by NIH in NIH Data Sharing Policy and Implementation Guidance and more specifically in "Data Sharing Expectations for National Institute of Mental Health (NIMH)-funded Clinical Trials". The data generated in this clinical trial will be entered into the NIMH Data Archive repository, as required by the Notice of Award, and presented at national and international conferences and published in a timely fashion. All final peer-reviewed manuscripts that arise from this trial will be submitted to the digital archive PubMed Central. Published data will be available in print or electronically from publishers, subject to subscription or printing charges. Research data that document, support and validate research findings will be made available after the main findings from the final research data set have been published.
Time Frame: 6 months after publication of study results

REFERENCES:
- [Background] Betancourt TS, McBain R, Newnham EA, Akinsulure-Smith AM, Brennan RT, Weisz JR, Hansen NB. A behavioral intervention for war-affected youth in Sierra Leone: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2014 Dec;53(12):1288-97. doi: 10.1016/j.jaac.2014.09.011. Epub 2014 Oct 2. PMID 25457927
- [Derived] Desrosiers A, Carrol B, Ritsema H, Higgins W, Momoh F, Betancourt TS. Advancing sustainable implementation of an evidence-based mental health intervention in Sierra Leone's schools: protocol for a hybrid type 3 implementation-effectiveness trial. BMC Public Health. 2024 Feb 3;24(1):362. doi: 10.1186/s12889-024-17928-w. PMID 38310232